CLINICAL TRIAL: NCT04303884
Title: Phase 2 Trial for Chemo-Resistant Gestational Trophoblastic Neoplasias With Pembrolizumab
Brief Title: Phase 2 Trial for Chemo-Resistant Gestational Trophoblastic Neoplasias With Pembrolizumab (CR-GTP)
Acronym: CR-GTP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CHA University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Min Chul Choi, Associate Professor, CHA University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pembro_CR-GTP
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Gestational Trophoblastic Neoplasia
Keywords: Gestational Trophoblastic Neoplasia; pembrolizumab; PD L1
MeSH Terms: conditions — Gestational Trophoblastic Disease | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Chemo-Resistant Gestational Trophoblastic neoplasias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: Pembrolizumab (Experimental): Chemo-resistant gestational trophoblastic neoplasias treated with pembrolizumab
  Interventions: Drug: Pembrolizumab Injection [Keytruda]

INTERVENTIONS:
Drug: Pembrolizumab Injection [Keytruda] — Pembrolizumab administration at a fix dose of 200 mg every 3 weeks

SUMMARY:
Gestational trophoblastic neoplasia (GTN) represents a group of rare tumors that accounts for less than 5% of gynecologic cancers which arising from malignant transformation of trophoblast, a cell originating from placenta. Placental expression of paternal antigens make placenta a target for maternal immune recognition during pregnancy, and PD-L1 expression maintains gestational tolerance. Also in GTN, PD-L1 is strongly expressed, suggesting the ligand is involved in tumor-immune evasion.

Most female patients with GTN cured with chemotherapy, however less than 5.0% of them die as a result of multi-drug resistance, necessitating novel approaches. Although there was limited data due to its rarity, the treatment response of avelumab and pembrolizumab in GTN is excellent (50% ~ 71.4% complete remission rate), as reported in the previous studies.

Therefore targeting of interaction PD-1/PD-L1 inhibition could be effective therapeutic strategy in chemoresistant GTN.

This study investigate clinical efficacy of patients with GTN resistant/refractory to multi-agent chemotherapy who treat with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of gestational trophoblastic neoplasia (hydatidiform-mole, invasive mole, gestational choriocarcinoma, placental site trophoblastic tumor, and epithelioid trophoblastic tumor) refractory or chemo-resistant to multi-agent chemotherapy (such as EMA-CO, EMA-EP, BEP, TP-TE etc.) status will be enrolled in this study.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
* Not a woman of childbearing potential
* The participant provides written informed consent for the trial.
* Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded tissue blocks are preferred to slides. It might be enrolled in this study even if tissue is not available for a variety of reasons.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation.
* Have adequate organ function as defined in the followings;

  1. Patients with adequate bone marrow function measured within 28 days prior to administration of study treatment as defined below : Absolute granulocyte count ≥ 1.5 x 10 9 /L ; Platelet count ≥ 100 x 10 9 /L ; Haemoglobin ≥ 9.0 g/dL (may have been blood transfused)
  2. Patients with adequate renal function : Calculated creatinine clearance ≥ 30 ml/min according to the Cockcroft-Gault formula (or local institutional standard method)
  3. Patients with adequate hepatic function : Serum bilirubin ≤ 1.5 x UNL and AST/ALT ≤ 2.5 X UNL (≤ 5 X UNL for patients with liver metastases)

Exclusion Criteria:

* GTN is a pregnancy-related tumor, all candidates will be positive for pregnancy test. Therefore, a positive pregnancy test is not exclusion criteria.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has a known history of Human Immunodeficiency Virus (HIV) infection.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Radiological response assessed by the overall response according to iRECIST criteria assessed by imaging (CT scan and/or MRI if contraindicated). | 12 months
Serologic response assessed by serum b-hCG | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Soo Im Park, RN, Study Director — CHA Bundang Medical Center
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided